CLINICAL TRIAL: NCT04923815
Title: A Real-world Study of Cardiac Ablation for Paroxysmal Supraventricular Tachycardia Using THERMOCOOL SMARTTOUCH® Diagnostic/Ablation Deflectable Tip Catheter（ST in PSVT-RWS）
Brief Title: A Real-world Study of Cardiac Ablation for PSVT Using ST Catheter
Acronym: ST in PSVT-RWS
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Medical (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BWI_2020_01
Record Dates: First submitted 2021-04-29; First posted 2021-06-11 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: AVRT, AVNRT
Keywords: AVRT, AVNRT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- AVNRT: atrioventricular nodal reentrant tachycardia
  Interventions: Device: THERMOCOOL SMARTTOUCH® Diagnostic/Ablation Deflectable Tip Catheter
- AVRT: atrioventricular reentrant tachycardia, including Wolff-Parkinson-White syndrome（WPW）
  Interventions: Device: THERMOCOOL SMARTTOUCH® Diagnostic/Ablation Deflectable Tip Catheter

INTERVENTIONS:
Device: THERMOCOOL SMARTTOUCH® Diagnostic/Ablation Deflectable Tip Catheter — THERMOCOOL SMARTTOUCH® catheter is a pressure catheter irrigated with cold saline, contact force sensing catheter. When used with Carto ®3 system, this catheter can provide a real time measurement for contact force. The magnitude and direction of the contact force can be displayed visually in the form of vector arrow on the top of catheter in Carto®3 system. It can be used for electrophysiological mapping and ablation of the heart.

SUMMARY:
Paroxysmal supraventricular tachycardia known as PSVT includes atrioventricular reentrant tachycardia (AVRT) and atrioventricular nodal reentrant tachycardia (AVNRT).

This study is multicenter, retrospective, cohort study. This study will collect real world data of AVNRT and AVRT cohorts retrospectively to evaluate the effectiveness and safety in real world clinical practice. 300 subjects with PSVT will be consecutively enrolled backwards since 02 Nov 2017, and at least 100 subjects for each cohort.

Cohort one: AVNRT Cohort two: AVRT, including Wolff-Parkinson-White syndrome（WPW）

ELIGIBILITY:
Inclusion Criteria:

1. Waiver of informed consent is approved by Ethics Committee, or follow methods approved by Ethics Committee to get patient's informed consent (such as get informed consent by telephone contact, etc.).
2. Patients diagnosed as atrioventricular reentrant tachycardia (AVRT), atrioventricular node reentrant tachycardia (AVNRT) after surgery/discharge, and the existing source records must include 1) at least 1 copy of preoperative ECG or intraoperative electrophysiological examination results;2) Information about the acute procedure outcome.
3. Patients were ablated by ST catheter.
4. Adult patients 18 years or older.

Exclusion Criteria:

1. Contraindications for the use of ST catheters, including:

   1. Ventriculotomy or atriotomy was performed within 8 weeks before the procedure;
   2. Presence of myxoma or intracardiac thrombus;
   3. fitted with artificial valves;
   4. Active systemic infection;
   5. Atrial septal patch.
2. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients with PSVT who meet eligibility criteria and were ablated with ST catheters will be consecutively enrolled backwards since 02 Nov 2017. Two cohorts are atrioventricular reentrant tachycardia (AVRT) and atrioventricular nodal reentrant tachycardia (AVNRT). Each of them contains at least 100 subjects.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Acute success rate of PSVT ablation using ST Catheter | Intra-procedure
  Acute success rate is defined as accessory pathway/slow pathway blockade immediately after ablation, and drug and/or electrophysiological stimulation no longer induces clinical arrhythmias.
Incidence of primary adverse events (PAE) | From procedure to pre-discharge (an average of 2-3 days)
  Primary adverse events include device or procedure related death, myocardial infarction, atrioventricular block, thrombosis, stroke/cerebral vascular accidents (CVA), tamponade/perforation, transient ischemia attack (TIA), pericarditis, major vascular complications/bleeding, Adverse Event which prolonged hospitalization due to non-arrhythmic causes.

SECONDARY OUTCOMES:
Acute success rate of cardiac ablation for AVNRT using ST catheter | Intra-procedure
  defined as accessory pathway blockade, and clinical arrhythmia could not be induced by drug and/or stimulation.
Acute success rate of cardiac ablation for AVRT using ST catheter | Intra-procedure
  defined as slow pathway blockade, and clinical arrhythmia could not be induced by drug and/or stimulation.
The proportion of patients who did not develop PSVT recurrence | from discharge to the follow-up visit (an average of 4-6 years)
  Data can be collected from hospital medical records/database and Telephone Survey Questionnaire. Recurrence of PSVT includes recurrence of PSVT identified by electrocardiogram or other cardio-electrical equipment, re-admission due to PSVT, re-procedure due to PSVT, take anti-arrhythmic drug due to PSVT, suffering typical PSVT symptoms.
Incidence of serious adverse events | from discharge to the follow-up visit (an average of 4-6 years)
  Data can be collected from hospital medical records/database and Telephone Survey Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Professor, Principal Investigator — Beijing Anzhen Hospital; Haixiong Wang, Professor, Principal Investigator — Shanxi Cardiovascular Hospital; Shanglang Cai, Professor, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (3):
- China (3):
  - Beijing Anzhen hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.